CLINICAL TRIAL: NCT00128362
Title: Clinical Trial of Sentinel Node Biopsy Versus Axillary Sampling in Women With Clinically Node Negative Operable Breast Cancer
Brief Title: Sentinel Node Biopsy and Axillary Sampling in Operable Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After initiation of study many studies reported an equivalence of SNB and ALND which led to widespread adoption of the former as standard procedure.
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TMH/115/2003; No.5/13/66/2003-NCD-III
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Cancer of the Breast
Keywords: Sentinel node; Axillary sampling; Operable breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Radio guided Sentinle node biopsy (Experimental): The radiolabeled Tc-99 colloid or phytate (500 Mbq) will be injected into the primary tumor 2 hours before surgery. A localized scintiscan will then be performed to confirm the radiolabeling of the sentinel node before surgery and for documentation. Isosulphan blue dye will be injected subdermal (0.5ml) over the tumor and intraparenchymal (3-4ml) towards the axilla 10-15mins before incision.
  Interventions: Procedure: Radio-guided sentinel node biopsy; Procedure: Axillary sampling

INTERVENTIONS:
Procedure: Radio-guided sentinel node biopsy
Procedure: Axillary sampling

SUMMARY:
The advent of mammography and increased awareness of breast cancer has resulted in detection of smaller tumors, the majority of which would not have had metastasized to the axillary lymph nodes. The sentinel node (SN) is presumably the first echelon node in the axillary basin to become involved with metastatic breast cancer cells. Sentinel node biopsy (SNB) in operable breast cancer has gained popularity since it promises to avoid treatment of the axilla when the nodes are negative for metastasis. Advances in technology (radio-guided SNB) is associated with a risk of false negative SN reporting in 4-12%. The consequence of leaving behind untreated positive non-sentinel nodes in the axilla is a potential risk for axillary recurrence. Axillary sampling is a simple and inexpensive procedure in which level I nodes are removed by a blind dissection. The investigators critically analyzed the efficacy of both the procedures separately in consecutive pilot studies i.e., targeted SNB versus blind axillary sampling. The current study is planned as a prospective comparison study where a patient undergoes both the procedures in the same surgical intervention and thus provides an immediate comparison of the two techniques with respect to their effectiveness.

DETAILED DESCRIPTION:
Axillary node dissection in operable breast cancer provides an accurate way of staging the disease. With increased popularity of screening and earlier diagnosis, most women do not harbor axillary metastases, in which case, axillary lymph node dissection could be avoided. Sentinel node biopsy (SNB) gained rapid popularity because the technique could predict the presence of metastases in downstream lymph nodes, so that surgery and its associated morbidity could be safely avoided. SNB can be performed with injection of isosulphan blue subdermally and peritumorally alone or in combination with radio-guidance with technetium-99 labeled colloid injection. Radio-guided SNB is superior to the blue dye in identifying the SN, and a combined technique is still better. However, it failed to accomplish its objective in a proportion of cases where the sentinel node could not be identified even with expensive gadgetry like gamma probes. An overview of sentinel node studies showed that the node was found in only 85-90% of patients and the overall sensitivity in correctly predicting the negative axilla by sentinel node biopsy was only 94%. There was a false negative rate of 6.2% wherein the sentinel node was reported negative in presence of metastasis to non-sentinel nodes in axilla.

Axillary sampling was a forerunner to the targeted sentinel node biopsy. The main objective of axillary sampling at that time was to detect a positive axilla. More recently it is being tested as an accurate predictor of axillary status for absence of metastasis.

There is a definite learning curve in SNB with higher non-detection rates and false negative rate in the earlier phases of the study compared to the later part. This learning curve is absent in axillary sampling, which requires no specialized training or expensive equipment and has a 100% detection rate. The mean number of sentinel nodes that were identified, as reported in various SNB studies, was 2.13 (with a range of mean numbers of SN dissected being 1.3-3.1). The actual range of number of sentinel nodes dissected was 1 - 8, which is quite comparable to the average 4 -5 nodes that are required to be sampled for accurately predicting the axilla. Badwe and Mittra have concluded that sentinel node biopsy is expensive and is driven by lure for technology and fashion, and has little advantage over axillary node sampling in predicting a negative axilla.

There is a validation study of lower axillary sampling versus total axillary clearance reported by Steele et al in 1985 with a sensitivity of 100% and an accuracy of 99.5%. The more recent validation study of 5-node axillary sampling compared to level I-II dissection was reported from Stockholm on 416 operable breast cancer patients. The noteworthy finding was that in this study node sampling had a 100% yield, 97.3% sensitivity and a negative predictive value of 98.5% with a false negative rate of 2.7% in predicting the axilla. The comparative figures for SNB in the world overview are 94% sensitivity, 97% negative predictive value and a false negative rate of 6.5%.

Preliminary studies of SNB and axillary sampling at TMH Sentinel node biopsy by Isosulphan blue injection was performed as a validation pilot study at the Breast unit in TMH between April 1999 to November 2000 in 100 women with clinically node negative operable breast cancer. SN was found in 77% cases with a false negative rate of 16.6% and sensitivity of 76.1%. The procedure had a negative predictive value of 90.4% cases in predicting the rest of the axilla. The number of sentinel nodes dissected was 1-6 with an average of 1.4.

Axillary sampling was subsequently performed as a pilot study between May 2001 to August 2002 in 97 women with a similar clinical stage as above. Nodes were found in all patients (100%) in level I with a false negative reporting in 11% cases, sensitivity of 88.9%, negative predictive value of 100% and an average of 4 nodes dissected (range from 1-9).

In developing countries with limited resources, it may not be feasible for every institution to acquire a gamma probe. Axillary sampling may thus be a comparably cheaper and practical alternative to SNB. Axillary sampling and sentinel node biopsy should, however, be compared with respect to the resultant morbidity and false negative rates before adopting either method as standard clinical practice.

The Nottingham group have recently published the results of a prospective study to find out the value of adding SNB to 4-node axillary sampling (4NAS) within the same patient. Two hundred patients were accrued and 4NAS was found to have a lower false negative rate compared to SNB. We propose to compare the two procedures in a clinical trial with a comparison of respective false negative rates and sensitivity as the immediate end points.

Methodology:

Eligible women will be recruited in the study after obtaining an informed consent and centrally registered at the Clinical Research Secretariat at the Tata Memorial Hospital, Mumbai.

The radiolabeled Tc-99 colloid or phytate (500 Mbq) will be injected into the primary tumor 2 hours before surgery. A localized scintiscan will then be performed to confirm the radiolabeling of the sentinel node before surgery and for documentation. Isosulphan blue dye will be injected subdermal (0.5ml) over the tumor and intraparenchymal (3-4ml) towards the axilla 10-15mins before incision.

Axillary sampling will be performed first. A 2 cm incision will be made in the middle third of the proposed axillary clearance incision below the axillary hairline. All axillary fat and tissue in an area of 2cm diameter will be dissected out. The anterior limit of dissection is the posterior border of pectoralis major, the posterior limit of dissection is the anterior border of latissimus dorsi muscle, upper limit of dissection is the intercostobrachial nerve, and base is serratus anterior muscle on lateral chest wall. In those cases that undergo a mastectomy, the tissue in the axillary tail will be identified first and then removed as specified above.

After completion of sampling procedure, the remaining axillary tissue will be checked for any other node showing a blue discoloration or radioactivity and the same will be documented as found outside of axillary sampling. Axillary clearance will then be separately completed in all patients by standard technique after extending the incision without waiting for the frozen section report.

ELIGIBILITY:
Inclusion Criteria:

* Clinically node negative operable breast cancer
* No prior incision or excision biopsy

Exclusion Criteria:

* Palpable axillary lymph nodes
* Contraindications for injecting radiocolloid

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of methodologies in predicting status of axillary lymph nodes | Within 30 days after surgery
  The patient enrolled on this study will be planned for surgery and outcome will be measured after avability of histo-pathological report.

SECONDARY OUTCOMES:
Number of lymph nodes identified by sentinel node biopsy and axillary sampling | Within 30 days of surgery
  The patient enrolled on this study will be planned for surgery and outcome will be measured after avability of histo-pathological report.
Number of times the sentinel node is found within the sampled nodes | Within 30 days of surgery
  The patient enrolled on this study will be planned for surgery and outcome will be measured after avability of histo-pathological report.
False negative rate by each method | within 30 days of surgery
  The patient enrolled on this study will be planned for surgery and outcome will be measured after avability of histo-pathological report.
Negative predictive value for each method | within 30 days of surgery
  The patient enrolled on this study will be planned for surgery and outcome will be measured after avability of histo-pathological report.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, M.S., Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Badwe RA, Thorat MA, Parmar VV. Sentinel-node biopsy in breast cancer. N Engl J Med. 2003 Nov 13;349(20):1968-71; author reply 1968-71. doi: 10.1056/NEJM200311133492017. No abstract available. PMID 14614174
- [Derived] Parmar V, Hawaldar R, Nair NS, Shet T, Vanmali V, Desai S, Gupta S, Rangrajan V, Mittra I, Badwe RA. Sentinel node biopsy versus low axillary sampling in women with clinically node negative operable breast cancer. Breast. 2013 Dec;22(6):1081-6. doi: 10.1016/j.breast.2013.06.006. Epub 2013 Aug 13. PMID 23948301